CLINICAL TRIAL: NCT02012257
Title: Success Rate of Anterior Middle Superior Alveolar (AMSA) Nerve Block in Three Different Sites of Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ali Shokraneh, DDS, MS, Ali Shokraneh, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 2952
Record Dates: First submitted 2013-12-08; First posted 2013-12-16 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Anesthesia; Functional
Keywords: anterior middle superior alveolar nerve; electric pulp tester; local anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Anterior Site (Experimental): AMSA nerve block injection
  Interventions: Procedure: AMSA nerve block injectio
- Common Site (Experimental): AMSA nerve block injection
  Interventions: Procedure: AMSA nerve block injectio
- Posterior Site (Experimental): AMSA nerve block injection
  Interventions: Procedure: AMSA nerve block injectio

INTERVENTIONS:
Procedure: AMSA nerve block injectio — Sites of injection

SUMMARY:
AMSA nerve block injection is targeted anterior superior alveolar nerve and middle superior alveolar nerve branches of infraorbital nerve through nutrient canals. Therefore, central to second premolar teeth of one quadrant can be anesthetized. The aim of the present study was to evaluate the efficacy of AMSA nerve block injection at an anterior and a posterior positions compared to commonly administrated site.

DETAILED DESCRIPTION:
AMSA: Anterior middle superior alveolar

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject
* Subjects had all their maxillary teeth from second premolar of one side to the second premolar of another Neither of these teeth was non vital, nor had large restorations, prosthetic crowns, caries, periodontal disease, history of trauma, and hypersensitivity.

Exclusion Criteria:

* Use medications alleviating or altering the pain sensation
* Allergy to anesthetics Pregnancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Pulpal anesthesia of central incisor to second premolar by electric pulp tester (EPT) | After each injection (base line) to 60 minutes
  Each teeth were evaluated by electric pulp tester immediately after injection to 60 minutes every six minutes. Having no reaction to the EPT was the criterion of considering a tooth has been anaesthetized. Anesthesia was considered successful if no reaction to the maximum output for two consecutive tests.

CONTACTS AND LOCATIONS:
Overall Officials: Masoud Yaghmaei, DMD, MS, Study Chair — Shahid Beheshti University of Medical Sciences